CLINICAL TRIAL: NCT05795517
Title: A Phase 2 ,Multicentre, Randomised, Double Blind Double Simulation, Placebo and Positive Controlled Study to Evaluate the Efficacy and Safety of HSK31679 in Patients With Hypercholesterolemia With Non-alcoholic Fatty Liver Disease
Brief Title: Study of HSK31679 in Subjects With Hypercholesterolemia With Nonalcoholic Fatty Liver Disease（NAFLD）
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK31679-201
Record Dates: First submitted 2023-03-09; First posted 2023-04-03 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia; non-alcoholic fatty liver disease(NAFLD); THR-β
MeSH Terms: conditions — Hypercholesterolemia; Non-alcoholic Fatty Liver Disease | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- HSK31679 low dose (Experimental)
  Interventions: Drug: HSK31679 low dose
- HSK31679 medium dose (Experimental)
  Interventions: Drug: HSK31679 medium dose
- HSK31679 high dose (Experimental)
  Interventions: Drug: HSK31679 high dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Ezetimibe (Active Comparator)
  Interventions: Drug: Ezetimibe 10mg

INTERVENTIONS:
Drug: HSK31679 low dose — HSK31679 low dose and placebo of HSK31679 ，QD，oral，Day1 to week 12
  Arms: HSK31679 low dose
Drug: HSK31679 medium dose — HSK31679 medium dose and placebo of HSK31679 ，QD，oral，Day1 to week 12
  Arms: HSK31679 medium dose
Drug: HSK31679 high dose — HSK31679 high dose and placebo of HSK31679 ，QD，oral，Day1 to week 12
  Arms: HSK31679 high dose
Drug: Placebo — placebo ，QD，oral，Day1 to week 12
  Arms: Placebo
Drug: Ezetimibe 10mg — Ezetimibe 10mg+placebo of HSK31679 ，QD，oral，Day1 to week 12
  Arms: Ezetimibe

SUMMARY:
The purpose of this study is to assess the efficacy and safety of HSK31679 tablets compared with placebo in reducing low-density lipoprotein cholesterol (LDL-C) and MRI-PDFF after 12 weeks of treatment in patients with hypercholesterolemia and non-alcoholic fatty liver disease (NAFLD).

ELIGIBILITY:
Inclusion Criteria:

1. Must be willing to participate in the study and provide written informed consent.
2. Male or female aged 18 ≤ age < 65 at the time of signing the informed consent.
3. At the time of screening, patients who had not received lipid-regulation therapy within 6 weeks had fasting LDL-C≥3.34mmol/L（130mg/dL）.
4. (BMI) ≥18kg/m2 and female subjects ≥45.0 kg and male subjects ≥50.0 kg.
5. During screening, fasting triglyceride (TG) <5.65 mmol/L.
6. During screening,MRI-PDFF≥8%.
7. Weight changes≤5% in the 4 weeks prior to screening.

Exclusion Criteria:

1. Did not discontinue any lipid-regulating therapy or any drug or supplement that may affect lipid levels 6 weeks before randomization or is expected to do so during the study period.
2. Homozygous familial hypercholesterolemia (HoFH) was diagnosed by genetic or clinical criteria.
3. Dyslipidemia caused by other diseases or drugs, such as rheumatoid arthritis, nephrotic syndrome, Cushing's syndrome, hypothyroidism, renal failure, systemic lupus erythematosus, glycogen accumulation, myeloma, lipodystrophy, acute porphyria, polycystic ovarian syndrome, etc
4. Before screening, LDL-C plasma exchange was performed within 12 months.
5. In the past, PCSK9 inhibitors, Lomitapide and Mipomersen were used for treatment.
6. uncontrolled hypertension had systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg at screening/baseline.
7. type 1 diabetes, or newly diagnosed type 2 diabetes within 1 month, or poorly controlled type 2 diabetes, or who could not maintain the same hypoglycemic regimen during the study.
8. Stroke or transient ischemic attack (TIA), acute coronary syndrome, stable angina attack, severe deep vein thrombosis, or pulmonary embolism occurred in the 12 months prior to screening.
9. Major surgery (including but not limited to: coronary or other revascularization, coronary artery bypass surgery, and transplantation) within 12 months prior to screening or planned during the study period.
10. Chronic systemic disease or history, including but not limited to

    1. Have a serious cardiopulmonary disease or history,Neurological disease or history,Autoimmune disease,Chronic digestive disease or history
    2. Have thyroid disease or symptomatic abnormalities in thyroid function tests (e.g., thyroid stimulating hormone (TSH) < 1.0 x lower limit of normal (LLN) or > 1.5 x upper limit of normal (ULN))
    3. History of malignancy (excluding cured basal cell carcinoma of the skin, carcinoma in situ, and papillary thyroid carcinoma) or history of antitumor therapy within 5 years prior to screening
    4. Disease or medical history assessed by the investigator as likely to affect the study
11. Bariatric surgery within 12 months at the time of screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Percentage change in LDL-C from baseline at 12 week; | Baseline and Week 12
  Percentage change in fasting low-density lipoprotein cholesterol (LDL-C) from baseline after 12 weeks of treatment;
Percentage change in MRI-PDFF from baseline at 12 week； | Baseline and Week 12
  Percentage change of MRI-PDFF(change in liver fat content by nuclear magnetic resonance - Proton Density Fat Fraction) from baseline after 12 weeks of treatment;

SECONDARY OUTCOMES:
Percentage change in fasting LDL-C from baseline; | Week2,4,8
  Percentage change in fasting low-density lipoprotein cholesterol (LDL-C) from baseline after 2, 4, and 8 weeks of treatment;
The proportion of patients with MRI-PDFF decreased by > 30% | Baseline and Week 12
  After 12 weeks of treatment, the proportion of patients with MRI-PDFF decreased by > 30%;
Proportion of patients with LDL-C<3.34mmol/L（<130mg/dL） | Baseline and Week 12
  After 12 weeks of treatment, the proportion of patients with LDL-C<3.34mmol/L（<130mg/dL）
Percentage change of fasting TG from baseline; | Week2,4,8,12
  After 2, 4, 8, 12 weeks of treatment, Percentage change of fasting triglycerides (TG), from baseline;
Percentage change of fasting TC from baseline; | Week2,4,8,12
  After 2, 4, 8, 12 weeks of treatment, Percentage change of fasting total cholesterol (TC) from baseline;
Percentage change of fasting HDL-C from baseline; | Week2,4,8,12
  After 2, 4, 8, 12 weeks of treatment, Percentage change of fasting high-density lipoprotein cholesterol (HDL-C) from baseline;
Percentage change in body weight from baseline | Baseline and Week 12
  Percentage change in body weight from baseline after 12 weeks of treatment.
AUC0-τ of HSK31679 (All subjects) | up to 2,4,7 weeks
Cmax of HSK31679 (All subjects) | up to 2,4,7 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tsinghua Changgung Hospital, Tsinghua University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xue F, Ma W, Gao J, Chen J, Yue W, Bu P, Chen Q, Chen H, Sheng J, Chen L, Liu F, Li G, Zhu C, Zhong B, Zhang J, Cai Q, Wang L, Chen Y, Pei Z, Yao L, Lv L, Gao Y, Xia B, Ji X, Liu Y, Du L, Ma G, Hao K, Li F, Wu T, Huo Y, Wei L. Efficacy and Safety of HSK31679 in Asian Patients With MASLD: A Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2025 Aug 20:S1542-3565(25)00703-7. doi: 10.1016/j.cgh.2025.08.009. Online ahead of print. PMID 40846146